CLINICAL TRIAL: NCT04667637
Title: Improving Neuroprotective Strategy for Ischemic Stroke With Sufficient Recanalization After Thrombectomy by Edaravone Dexborneol (INSIST-ED): a Prospective, Randomized, Double Blinded, Multi-centre Study
Brief Title: Improving Neuroprotective Strategy for Ischemic Stroke With Sufficient Recanalization After Thrombectomy by Edaravone Dexborneol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hui-Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y(2020)045
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Stroke; Endovascular Thrombectomy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.9% NaCl (Placebo Comparator): Intravenous injections of 0.9% NaCl BID for 12 ±2days.
  Interventions: Drug: edaravone dexborneol
- Edaravone Dexborneol (Experimental): Intravenous injections of edaravone dexborneol (37.5mg in 0·9% NaCl) BID for 12 ±2days.
  Interventions: Drug: edaravone dexborneol

INTERVENTIONS:
Drug: edaravone dexborneol — Intravenous injections of edaravone dexborneol (37.5mg, dissolved in 100ml saline) twice a day for 12 ±2 days.
  Other Names: edaravone deborbeol placebo

SUMMARY:
To explore the safety and efficacy of edaravone dexborneol for the treatment of acute ischemic stroke patients who received endovascular thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age;
2. Patients who presented with acute ischemic stroke and a large vessel occlusion in the anterior circulation and met the criteria of mechanical thrombectomy;
3. Sufficient recanalization within 9 hours of stroke onset;
4. Sufficient recanalization （TICI 2b-3）;
5. Acute ischemic stroke with neurological baseline deficit equivalent to the National Institute of Health Stroke Scale (NIHSS) ≥ 6 before recanalization treatment;
6. First ever stroke or mRS≤1 after previous disease
7. The availability of informed consent.

Exclusion Criteria:

1. Acute ischemic stroke patients with insufficient recanalization（TICI < 2a）
2. Hemorrhagic transformation (PH2) indicated by NCCT performed after the operation immediately;
3. Hemorrhagic stroke: cerebral hemorrhage, subarachnoid hemorrhage;
4. Coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia （ <100000/mm3）;
5. Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
6. Severe hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg);
7. Patients with malignant tumor or under antineoplastic therapy with estimated lifetime less than 3 months;
8. Pregnancy, plan to get pregnant or during lactation;
9. Patients with contraindication or allergic to any ingredient of drugs in our study;
10. Unsuitable for this clinical studies assessed by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 2 | Day 90
  Proportion of patients with modified Rankin Score 0 to 2

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 1 | Day 90
  Proportion of patients with modified Rankin Score 0 to 1
Distribution of modified Rankin Score | Day 90
  Distribution of modified Rankin Score after the treatment
Changes in National Institute of Health stroke scale (NIHSS) | 24 hours, 48 hours, and 2 weeks
  the minimum and maximum values of NIHSS are 42 and 0, respectively; higher NIHSS mean a worse outcome
Change in infarct volume | 1 week
  infarct volume is determinted by CT or DWI

OTHER OUTCOMES:
Proportion of symptomatic intracranial hemorrhage (sICH) | 48 hours
  sICH was defined as 4 or more increase in NIHSS caused by hemorrhage
Proportion of intraparenchymal hemorrhage (PH1 and PH2) | 48 hours
  Proportion of PH1 and PH2 within 48 hours after the treatment
Proportion of death | Day 90
  death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen HS, Zhao ZA, Shen XY, Qiu SQ, Cui Y, Qiu J, Li W, Zhang H, Chen WH, Wang LH, Zhang DH, Chen Y, Ma YT, Gao ZE, Wang SC, Li D, Liu H, Nguyen TN. Edaravone dexborneol for ischemic stroke with sufficient recanalization after thrombectomy: a randomized phase II trial. Nat Commun. 2025 Mar 10;16(1):2393. doi: 10.1038/s41467-025-57774-x. PMID 40064868